CLINICAL TRIAL: NCT00580502
Title: A Prospective Study to Evaluate the Safety and Efficacy of LAP-BAND® Adjustable Gastric Band (LAGB®) Operations for Patients With BMI Between 30-40 kg/m2 With Co-morbidities
Brief Title: Safety and Efficacy of Adjustable Gastric Band Operations for Patients With Body Mass Index (BMI) Between 30-40 kg/m2
Acronym: LBMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Heekoung A Youn, Research coordinator, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H # 10686; 10686 (Other: NYULMC IRB); G030190 (Other: FDA)
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Obesity, 50 lbs overweight
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAGB for low BMI patients (Experimental): the LAP-BAND® Adjustable Gastric Band (LAGB®) for patients with BMI between 30-40 kg/m2 with co-morbidities
  Interventions: Device: LAP-BAND® Adjustable Gastric Band (LAGB®)

INTERVENTIONS:
Device: LAP-BAND® Adjustable Gastric Band (LAGB®) — Bariatric surgery for patient whose BMI is between 30 and 40 kg/m^2

SUMMARY:
This study is to evaluate the safety and efficacy of Gastric Banding for patients with body mass index (BMI) between 30-40 kg/m2 with medical conditions related to obesity.

DETAILED DESCRIPTION:
TITLE OF STUDY:A prospective study to evaluate the safety and efficacy of LAP-BAND® Adjustable Gastric Band (LAGB®) operations for patients with BMI between 30-40 kg/m2 with co-morbidities

CLINICAL PHASE: Phase III new indication for use of the device not yet approved by FDA

STUDY OBJECTIVES

* To determine the safety and efficacy of the LAP-BAND® Adjustable Gastric Band (LAGB®) for patients with BMI between 30-40 kg/m2 with co-morbidities
* To determine long-term effects on patients' co-morbidities

STUDY VARIABLES: Morbidity & mortality, percent of excess weight loss, nutritional status, improvement of pre-operative co-morbidities, weight loss maintained, and quality of life evaluation

DESIGN: Prospective single center study

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 and equal to or less than 60 years of age.
* BMI of at least 30 and maximum BMI of 40 with co-morbidities
* Willingness to comply with dietary restrictions required by the protocol
* History of obesity for at least 5 years
* History of at least 6 months of documented failures with traditional non-surgical weight loss methods
* Willingness to follow protocol requirements
* If female with childbearing potential, using an appropriate form of contraception

Exclusion Criteria:

* Age less than 18, age greater than 60
* Pregnancy
* History of major depressive disorder or psychosis
* Previous bariatric surgery or previous gastric surgery
* Presence of achalasia
* Presence of portal hypertension, cirrhosis, and/or varices
* Patient with inflammatory disease of the gastrointestinal tract such as Crohn's Disease
* Patients with autoimmune connective tissue disorders
* Patients with acute abdominal infections
* Any condition that, in the judgment of the investigator, would place a subject at undue risk, or potentially compromise the results or interpretation of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ren-Fielding, M.D., Principal Investigator — NYUSOM

REFERENCES:
- See also: NYU Program for Surgical Weight Loss — http://nyuweightloss.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Lap-Band: Low BMI patients who will go through Lap-band surgery.
  LAP-BAND® Adjustable Gastric Band (LAGB®): Bariatric surgery: LAGB
Period: Overall Study
Arm/Group | Lap-Band
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- LAP-BAND® Adjustable Gastric Band (LAGB®) Operations: A prospective study to evaluate the safety and efficacy of LAP-BAND® Adjustable Gastric Band (LAGB®) operations for patients with BMI between 30-40 kg/m2 with co-morbidities
Arm/Group | LAP-BAND® Adjustable Gastric Band (LAGB®) Operations
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 5
BMI [Mean (Standard Deviation); unit: kg/m2] | 35.1 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: To Determine Percent of Excess Weight Loss (%EWL) After Laparoscopic Adjustable Gastric Banding Surgery
Description: Change in weight from baseline at 5 years by calculating the percentage of the weight loss from the total excess weight.
Time Frame: 5 years
Population: All participants who underwent LAGB are included in the analysis population.
Measure: Mean (Standard Deviation); unit: percentage of excess weight loss
Groups:
- LAGB: LAGB surgery for the patient whose BMI between 30 and 40 kg/m^2
Arm/Group | LAGB
Number analyzed (Participants) | 46
percentage of excess weight loss | 51.74 (27.36)

2. Secondary Outcome: Level of LDL (Bad Cholesterol) After Laparoscopic Adjustable Gastric Band Surgery
Description: Change in level of LDL from baseline at 5 years
Time Frame: 5 years
Population: All participants who underwent LAGB are included in the analysis population.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | LAGB
Number analyzed (Participants) | 46
mg/dl | 117 (34)

3. Secondary Outcome: Level of Triglycerides (Bad Cholesterol) After Laparoscopic Adjustable Gastric Band Surgery
Description: Change in level of Triglycerides from baseline at 5 years
Time Frame: 5 years
Population: All participants who underwent LAGB and had 5 year follow up visit are included in the analysis population.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | LAGB
Number analyzed (Participants) | 46
mg/dl | 103 (58)

4. Secondary Outcome: Level of HbA1c (Blood Test for Diabetes) After Laparoscopic Adjustable Gastric Band Surgery
Description: Change in level of HbA1c from baseline at 5 years
Time Frame: 5 years
Population: All participants who underwent LAGB and had 5 year f/u visit are included in the analysis population.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | LAGB
Number analyzed (Participants) | 46
percentage of HbA1c | 5.6 (0.6)

ADVERSE EVENTS:
Time Frame: Entire 5 years study period
Arm/Group | LAP-BAND® Adjustable Gastric Band (LAGB®) Operations
Serious Adverse Events (participants affected / at risk) | 14/50
Other Adverse Events (participants affected / at risk) | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND® Adjustable Gastric Band (LAGB®) Operations (N=50)
Band revision/replacement (Surgical and medical procedures) | 14 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAP-BAND® Adjustable Gastric Band (LAGB®) Operations (N=50)
Port revision/replacement (Surgical and medical procedures) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No